CLINICAL TRIAL: NCT01585753
Title: Maraviroc Switch Vascular Endothelium (VE) Substudy: a Substudy of MARCH
Brief Title: MARCH Vascular Endothelium Substudy
Acronym: MARCH VE
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: MARCH-Kirby VE substudy
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular function; maraviroc
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Maraviroc

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Arm 1: NRTI and PI
  Interventions: Drug: NRTI + PI
- Arm 2: Maraviroc + PI
  Interventions: Drug: maraviroc + PI
- Arm 3: maraviroc + NRTI
  Interventions: Drug: maraviroc + NRTI

INTERVENTIONS:
Drug: NRTI + PI — tenofovir zidovudine abacavir lamivudine emtricitabine ritonavir darunavir atazanavir lopinavir fosamprenavir
  Groups: Arm 1
Drug: maraviroc + PI — maraviroc ritonavir darunavir atazanavir lopinavir fosamprenavir
  Groups: Arm 2
Drug: maraviroc + NRTI — maraviroc tenofovir zidovudine abacavir lamivudine emtricitabine
  Groups: Arm 3

SUMMARY:
This is a substudy of MARCH, in which we are exploring the changes in the vascular endothelium using pulse wave tonometry (a non invasive measure of cardiac health) to measure the changes in small and large arterial elasticity in participants of the MARCH study who switch to maraviroc-based regimens over 96 weeks of follow-up.

DETAILED DESCRIPTION:
Cardiovascular disease is increasingly recognised as a complication of HIV +/- therapies to treat it. Blood vessel elasticity, or compliance, can be depicted as the ability of the vessels to convert intermittent blood flow (cardiac ejection during systole) to continuous blood flow throughout the cardiac cycle. The compliance, or ability of vessels to accept energy, can be subdivided into elasticity of large and small vessels. Pulse wave tonometry is a non-invasive technique performed using a hand-held tonometer that generates two indices which correspond to large artery elasticity (LAE) and small artery elasticity (SAE). LAE and SAE estimates by pulse waveform analysis have previously shown greater correlation to Framingham risk when directly compared with other techniques such as flow-mediated diltation, and both LAE and SAE are associated with traditional cardiovascular risk factors (smoking, insulin resistance, hypertension).

It is unclear what the net effect of maraviroc, a chemokine-receptor blocker is on cardiovascular function.

The aims of this substudy are:

* To compare changes in the vascular endothelium between the control arm ((N(t)RTI) plus PI/r) and each of the maraviroc switch arms over 48 weeks of follow-up.
* To compare the changes in biomarkers and selected immunological markers between the control arm ((N(t)RTI) plus PI/r) and each of the maraviroc switch arms over 48 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled prior to treatment in the parent study;
* Provision of written, informed consent for participation in the substudy

Exclusion Criteria:

* Known supraventricular tachycardia such as atrial flutter and/or fibrillation that precludes the measurement of pulse wave using tonometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in MARCH
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean change in small arterial elasticity (SAE) as measure by pulse wave tonometry | 96 weeks
  measured at 6 timepoints week 0, 4, 12, 24, 48, 96

SECONDARY OUTCOMES:
• Mean change in large arterial elasticity (LAE) as measure by pulse wave tonometry | 96 weeks
  measured at 6 timepoints, week 0,4,12,24,48,96
• Changes from baseline in selected soluble markers of immune activation, coagulation, vascular and platelet function | 96 weeks
  stored bloods from the main study will be used to explore changes in vascular biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Pett, FRACP,FRCPE,PhD, Principal Investigator — Kirby Institute
Locations (6):
- Argentina (3):
  - Hospital General de Agudos "Dr. José María Ramos Mejía", Buenos Aires, Buenos Aires
  - Fundacion IDEAA, Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
- St. Vincent's Hospital, Sydney, New South Wales, Australia
- Johann Wolfgang Goethe-University Hospital, Medical HIVCENTER, Frankfurt, Frankfurt Am Main, Germany
- Chulalongkorn University Hospital, Bangkok, Bangkok, Thailand